CLINICAL TRIAL: NCT04175392
Title: Effect of Probiotics in Non-Alcoholic Fatty Liver Disease and Steatohepatitis Measured by Transient Elastography (PRONE Study).
Brief Title: Effect of Probiotics in Non-alcoholic Fatty Liver Disease and Steatohepatitis
Acronym: PRONE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Mariquit Sendelbach, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-129
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: Fatty Liver Disease; Fibrosis, Liver; Cirrhosis, Liver; Steatohepatitis, Nonalcoholic
Keywords: Fatty Liver; Fibrosis; Cirrhosis; Probiotic; Steatohepatitis; Elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fatty Liver; Fibrosis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind study. Participant will be randomized to either the Treatment (Probiotic) Group or the Control (Placebo) Group.
Who Masked: Participant, Investigator
Masking Description: Both Participants and Researchers will not know which treatment group assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group: Probiotic (Active Comparator): Probiotic 1 billion units Supplement Once Daily
  Interventions: Drug: Align Probiotic Supplement Capsule
- Control Group: Placebo (Placebo Comparator): Placebo Capsule Once Daily
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Align Probiotic Supplement Capsule — Align Probiotic 1 billion units, 1 capsule once daily
  Other Names: Probiotic
  Arms: Treatment Group: Probiotic
Drug: Placebos — Placebos capsule 1 capsule Once daily
  Other Names: Placebo
  Arms: Control Group: Placebo

SUMMARY:
This study will evaluate the effect of probiotics, a beneficial intestinal bacteria supplement, if it will cause improvement of the non-alcoholic fatty liver disease (NAFLD) and or non-alcoholic steatohepatitis (NASH- an inflammation with concurrent fatty accumulation of the liver) as measured by transient elastography - an ultrasound of the liver that assess the elastic properties (density) and stiffness of the liver tissue. This study will enroll patients 18 years and older with diagnosis of NAFLD and or NASH.

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) and Non-Alcoholic Steatohepatitis (NASH) are conditions without symptoms where inflammation in the liver can progress to end-stage liver disease (cirrhosis). Current standard of care for these conditions include control of metabolic syndrome which includes but is not limited to a patient's high blood pressure (hypertension), high cholesterol (hyperlipidemia), high blood sugar (hyperglycemia) and excess fat around the waist (central obesity and waist circumference) with lifestyle modifications including diet, exercise and medications. While the mechanism for inflammation on the liver in NAFLD and NASH is not completely understood, the American Association for the Study of Liver Diseases currently suspects it may be connected with the metabolism in the bowel and subsequent hepatic (liver) circulation. The bacteria of the intestines (microbiome or gut flora) may play a role in the inflammatory cascade through the bloodstream that affects the liver.

The World Health Organization (WHO) and the Food and Agricultural Organization (FAO) of the United Nations define Probiotics as a "live microorganism" which, when taken in adequate amounts confer a health benefit in the gastrointestinal tract. This study will be done to determine if probiotic use may be a viable treatment option for NAFLD and NASH and to establish a link that the intestinal microbiome or gut flora plays a role in liver inflammation which will be measured by elastography.

Patients with NAFLD and NASH seen in office consultation of the investigator will be approached to participate in the randomized like a flip of a coin, double-blind (patients and researchers will be blinded), placebo controlled study. Participant will be counseled on diet and exercise. The participants will receive information on a standardized Mediterranean diet based nutrition program as well as direction for recommended 30 minutes of aerobic exercise 3 times weekly. A baseline transient elastography, blood test such as liver enzymes Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) will be drawn, including hemoglobin A1C (diabetic marker), cholesterol in the form of Low-Density Lipoprotein (LDL/bad cholesterol) and assessment of Body Mass Index (BMI).

Participants will be randomized by pharmacy into 2 groups, a control group and a treatment group. The treatment group will be provided with a 6 month supply of Align probiotic once daily supplementation; the control group will be given a placebo for 6 months along with both groups given instructions on how to take the supplement. Subjects will receive a 1 month phone call follow up to ensure adherence to study instructions and daily oral intake of supplement, and again at 3 months. Study participation will end at 6 months after the repeat of liver enzymes, hemoglobin A1C, lipid panel, assessment of BMI and transient elastography as completed at scheduled clinical appointment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD and/or NASH
* Subject aged 18 and older
* Non-pregnant - Self-reported
* Subject with decision making capacity to understand and consent to study procedures
* Ability to follow study related activities regarding medications, diet and exercise

Exclusion Criteria:

* Without diagnosis of NAFLD or NASH
* History of liver disease from other causes, including but not limited to hepatitis, autoimmune, alcohol use, fatty liver of pregnancy, Wilson's disease, primary or secondary hemochromatosis
* Patients aged less than 18 years
* Self-reported pregnant patients
* Inability to understand, follow and consent to study procedures
* Hepatic decompensation defined as gastrointestinal bleeding, ascites, hepatic encephalopathy
* Inability to engage in exercise
* Currently immunocompromised or taking immunosuppressive drugs
* Milk protein allergy
* Recent or active chemotherapy for malignancy
* Gastrointestinal malignancy
* Gastrointestinal disease such as Ulcerative Colitis, Crohn's Disease as these alter the microbiome
* Recent antibiotic therapy (within 6 months)
* Known allergy to probiotics
* History of major gastrointestinal surgery such as resection of the colon
* No concomitant use of probiotic from any source (i.e., kefir, certain yogurts, live culture, sauerkraut)
* Liver scan >2 months prior to enrollment
* Weight loss >5 pounds in the last 2 months
* Any implanted battery operated device (i.e. AICD, pacemaker, loop recorder, cochlear implant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariquit Sendelbach, DO, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital, Farmington Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
Started | 7 | 7
Completed | 4 | 5
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Probiotic Effects on Liver Fibrosis
Description: Probiotic effects on liver fibrosis as measured by transient elastography, as a change from baseline to 6 months, measured on a scale from 1-4. 1= a clinical grade of F0-F1 and represents 2-7 kilopascals in elastography testing. 4= a clinical grade of F4 and represents 14 kilopascals or higher in elastography testing. A higher score on the scale represents worsening liver scarring. Positive numbers indicate an increase in fibrosis; negative numbers indicate decrease in fibrosis.
Time Frame: 6 months
Population: Only 1 participant in group 1 and 2 participants in group 2 completed the 6 month fibroscan. Data available only for these participants.
Measure: Mean (Standard Deviation); unit: units on a 1-4 scale
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
Number analyzed (Participants) | 1 | 2
units on a 1-4 scale | -1 (0) | 0 (0)

2. Secondary Outcome: Probiotic Effects on Liver Enzymes, AST
Description: Probiotic effects on Liver enzymes, AST as a change from baseline to 6 months, measured in units per liter. Positive numbers indicate an increase in AST; negative numbers indicate decrease in AST
Time Frame: 6 months
Population: 2 participants in the treatment group and 2 participants in the placebo group withdrew before 6 months: data not available for these 4 participants.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
Number analyzed (Participants) | 5 | 5
units per liter | -3.8 (15.0) | 4.0 (13.9)

3. Secondary Outcome: Probiotic Effects on Liver Enzymes, ALT
Description: Probiotic effects on Liver enzymes, ALT as a change from baseline to 6 months, measured in units per liter. Positive numbers indicate an increase in ALT; negative numbers indicate decrease in ALT
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
Number analyzed (Participants) | 5 | 5
units per liter | 2.2 (27.3) | -4.6 (26.3)

4. Secondary Outcome: Probiotic Effects on Diabetic Markers
Description: Probiotic effects on Diabetic Markers as measured by hemoglobin A1C blood test as a change from baseline to 6 months, measured in percent. Positive numbers indicate an increase in hemoglobin A1c; negative numbers indicate decrease in hemoglobin A1c
Time Frame: 6 months
Population: 4 participants in the control group and 3 participants in the placebo group did not have this test performed: data not available for these 7 participants.
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
Number analyzed (Participants) | 3 | 4
percentage of total hemoglobin | .63 (.5) | .15 (.2)

5. Secondary Outcome: Probiotic Effects on BMI
Description: Probiotic effects on Body Mass Index (BMI) wherein weight and height will be combined to report BMI in kg/m^2 as a change from baseline to 6 months. Positive numbers indicate an increase in BMI; negative numbers indicate decrease in BMI.
Time Frame: 6 months
Population: 4 participants in the control group and 2 participants in the placebo group did not have BMI completed at 6 months: data not available for these 6 participants.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
Number analyzed (Participants) | 3 | 5
kg/m^2 | -.26 (1.5) | -1.85 (2.6)

6. Secondary Outcome: Probiotic Effects on LDL
Description: Probiotic effects on Low-density Lipoprotein (LDL) as a change from baseline to 6 months, measured in milligrams per deciliter. Positive numbers indicate an increase in LDL; negative numbers indicate decrease in LDL
Time Frame: 6 months
Population: 4 participants in the treatment group and 4 participants in the placebo group did not have LDL completed at 6 months: data not available for these 8 participants.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
Number analyzed (Participants) | 3 | 3
milligrams per deciliter | -9.3 (32.4) | 29.75 (45.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment Group: Probiotic | Control Group: Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Probiotic (N=7) | Control Group: Placebo (N=7)
Increased gas (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT04175392/Prot_SAP_000.pdf